CLINICAL TRIAL: NCT04666714
Title: National, Multicentre, Randomized, Double-blind, Double-dummy Phase III Clinical Trial to Evaluate the Efficacy and Safety of Praga Formulation in the Treatment of Neuropathic Pain
Brief Title: Efficacy and Safety of Praga Formulation in the Treatment of Neuropathic Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1719 - PRAGA
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Praga formulation (Experimental): The study is double-dummy. The participant must take pills twice a day, as follows:
  Morning:Placebo pregabalin tablet, oral Night: Placebo pregabalin tablet, oral plus Praga formulation,oral
  Interventions: Drug: Praga formulation; Other: Placebo pregabalin 75mg; Other: Placebo Pregabalin 150mg
- Pregabalin (Active Comparator): The study is double-dummy. The participant must take pills twice a day, as follows:
  Morning:Pregabalin tablet, oral Night: Pregabalin tablet plus, oral placebo Praga formulation, oral
  Interventions: Drug: Pregabalin 75mg; Drug: Pregabalin 150mg; Other: Placebo Praga formulation

INTERVENTIONS:
Drug: Praga formulation — Praga formulation tablet
  Arms: Praga formulation
Other: Placebo pregabalin 75mg — Placebo pregabalin 75mg tablet
  Arms: Praga formulation
Other: Placebo Pregabalin 150mg — Placebo Pregabalin 150mg tablet
  Arms: Praga formulation
Drug: Pregabalin 75mg — Pregabalin 75mg tablet
  Arms: Pregabalin
Drug: Pregabalin 150mg — Pregabalin 150mg tablet
  Arms: Pregabalin
Other: Placebo Praga formulation — Placebo Praga formulation tablet
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Praga formulation in the treatment of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants of 18 years and older;
* Diagnosis of type 2 or type 1 diabetes for at least 1 year;
* No change in antidiabetic medication winthin 3 months;
* Diagnosis of painful sensorimotor diabetic polyneuropathy;
* Presence of at least one of the following symptoms: i. numbness in the toes, feet and / or legs; ii. paresthesias (tingling and / or neuropathic pain) in the toes, feet and / or legs.
* Presence of at least one of the following signs: i. symmetrical hypoesthesia of tactile, thermal or painful sensation (s) in the distal region of the legs; ii. hypoactive or abolished achilles reflexes;
* Glycated hemoglobin ≤ 11%;
* Score ≥ 12 points on the LANSS pain scale (Leeds Assessment of Neuropathic Symptoms and Signs); j) Participants with moderate to severe pain, a score ≥ 4 on the numerical pain scale (0-10 points);
* Participants with moderate to severe neuropathic pain who recorded in the diary a minimum of 4 of the 7 days from the period to assess the baseline pain score.

Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 2 years;
* Pregnant women, breastfeeding or planning to become pregnant, or women with the potential to become pregnant who are not using a reliable method of contraception;
* History of pernicious anemia, uncontrolled hypothyroidism, chronic hepatitis B;
* HIV diagnosis;
* History of neurological disorder unrelated to diabetic neuropathy;
* Non-responders to previous pregabalin treatment;
* High variability in the baseline pain score;
* Other conditions that may alter the sensitivity in the affected dermatome or in the area involved in neuropathic pain that may confuse pain assessment;
* Severe psychiatric condition;
* Cognitive decline that affect the participant from correctly answering the scales and questionnaires;
* Clinically relevant cardiac abnormalities, which at the researcher's discretion represent a risk to participation in the trial;
* Participant who has amputated lower limb due to complications from diabetes;
* Renal failure, defined by the estimated glomerular filtration rate [eGFR] <60 mL / min / 1.73 m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain intensity. | 3 months
  The change in pain intensity from baseline after 3 months of treatment will be scored by Numerical Rating Scale from 0 to 10 points, with 0 = no pain and 10 = worst possible pain, recorded in a participant diary.

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 6 months
  The incidence and severity of adverse events recorded during the study will be determined over 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Allegisa, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No